CLINICAL TRIAL: NCT03329885
Title: A Double-Blind Randomized Placebo-Controlled Single and Multiple Ascending Doses Study of the Safety and Tolerability, Pharmacokinetics (Including Bioavailability Comparison and Food Effect) and Pharmacodynamics of Oral BMS-986251 Administration in Healthy Subjects, With Efficacy Assessment of Multiple Doses in Patients With Moderate-to-Severe Psoriasis
Brief Title: A Study of Experimental Medication BMS-986251, Taken by Mouth, in Healthy Participants and Patients With Average to Very Serious Psoriasis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Adverse change in the risk/benefit
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM024-005; 2017-003408-38 (EudraCT Number)
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Results first posted 2019-10-21 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-09

CONDITIONS: Rheumatoid Arthritis; Psoriasis; Ankylosing Spondylitis; Inflammatory Bowel Diseases; Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Psoriasis; Spondylitis, Ankylosing; Inflammatory Bowel Diseases; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A Single Ascending Dose (SAD) in Healthy Patients (Experimental): Healthy patient will receive single escalating oral doses of BMS-986251 or placebo
  Interventions: Drug: BMS-986251; Other: Placebo
- Part B Multiple Ascending Dose (MAD) in Healthy Patients (Experimental): Healthy patients will receive daily escalating oral doses of BMS-986251 or placebo
  Interventions: Drug: BMS-986251; Other: Placebo
- Part C Multiple Dosing in Psoriasis Patients (Experimental): Psoriasis patients will receive daily escalating oral doses of BMS-986251 or placebo
  Interventions: Drug: BMS-986251; Other: Placebo

INTERVENTIONS:
Drug: BMS-986251 — Escalating oral dose
Other: Placebo — Escalating oral dose

SUMMARY:
The purpose of this study is to investigate experimental medication BMS-986251 taken by mouth in healthy patients and patients with average to very serious Psoriasis (a condition characterized by itchy, dry skin with a scaly rash).

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria (Healthy Patients):

* Males and females, ages 18 to 55 years, inclusive, at screening
* Healthy subjects, as determined by no clinically significant deviations from normal in medical history, physical examination, 12-lead ECGs, vital signs, and clinical laboratory results
* Body mass index (BMI) of 18.0 to 30.0 kg/m2, inclusive, at screening
* Body weight between 55 kg and 105 kg, inclusive, at screening
* Women must not be breastfeeding

Exclusion Criteria (Healthy Patients):

* Previous participation in the current study
* Participation in a drug study or exposure to any investigational drug or placebo within 2 months prior to (the first) drug administration in the current study
* Employees of PRA or the Sponsor and their relatives
* Any significant acute or chronic medical condition that presents a potential risk to the subject and/or that may compromise the objectives of the study, including active, or history of, liver disease, or intestinal disorder including irritable bowel syndrome
* Current or recent (within 3 months of study treatment administration) gastrointestinal disease that could affect pharmacokinetics; history of cholecystectomy is not allowed

Inclusion Criteria (Psoriasis Patients):

* Males and females, ages 18 to 70 years, inclusive, at screening
* BMI of 18.0 to 35.0 kg/m2, inclusive, at screening
* Body weight between 55 kg and 120 kg, inclusive, at screening
* Diagnosed with stable chronic plaque psoriasis, for at least 6 months prior to screening and be candidates for either photo-therapy or systemic treatment
* Moderate-to-severe intensity of psoriasis as defined by:

  1. Affected body surface area (BSA) of ≥10%
  2. Psoriasis Area and Severity Index (PASI) ≥12
  3. Physician Global Assessment (PGA; 6-point scale) ≥3

Exclusion Criteria (Psoriasis Patients):

* Previous participation in the current study
* Participation in a drug study or exposure to any investigational drug or placebo within 2 months prior to (the first) drug administration in the current study
* Employees of PRA or the Sponsor and their relatives
* Any significant acute or chronic medical condition that presents a potential risk to the subject and/or that may compromise the objectives of the study, including active, or history of, liver disease, or intestinal disorder including irritable bowel syndrome
* Current or recent (within 3 months of study treatment administration) gastrointestinal disease that could affect pharmacokinetics; history of cholecystectomy is not allowed

Other protocol defined inclusion/exclusion criteria could apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Groningen, Netherlands

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 96 participants were enrolled (screened) of whom 36 were screen failures, 22 were approved but not dosed and 38 were randomized in the study.
Groups:
- Part A: Placebo; Part A: BMS-986251 2 mg; Part A: BMS-986251 6 mg; Part A: BMS-986251 15 mg; Part A: BMS-986251 30 mg; Part A : BMS-986251 60 mg: Part A Single Ascending Dose (SAD) in Healthy Participants; single escalating oral doses of BMS-986251 or placebo
- Part B: Placebo; Part B: 3 mg QD (Once Daily): Part B Multiple Ascending Dose (MAD) in Healthy Participants; daily escalating oral doses of BMS-986251 or placebo
- Part C: Multiple Dosing in Psoriasis Patients: Psoriasis patients to receive daily escalating oral doses of BMS-986251 or placebo
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily) | Part C: Multiple Dosing in Psoriasis Patients
Started | 9 | 6 | 6 | 6 | 6 | 3 | 1 | 1 | 0 (Due to early termination of study, Part C was cancelled and no patients were dosed)
Completed | 9 | 6 | 6 | 6 | 6 | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Sponsor discontinued the study early | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All demographic characteristics for Part A are summarized. Due to early termination of the study, only 1 participant was enrolled in the placebo group and 1 participant in the BMS-986251 group in Part B. Part B demographics data is not reported for privacy reasons.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Total
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 3 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.9 (10.46) | 34.5 (7.96) | 32.3 (11.64) | 37.2 (12.26) | 33.8 (12.52) | 29.0 (6.56) | 33.1 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 2 | 3 | 3 | 0 | 18
  Male | 4 | 1 | 4 | 3 | 3 | 3 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 9 | 5 | 6 | 6 | 6 | 3 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 0 | 0 | 0 | 3
  White | 7 | 4 | 4 | 6 | 6 | 3 | 30
  More than one race | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced the Following: Serious Adverse Events (SAEs), Death or an Adverse Event (AE) Leading to Study Discontinuation
Description: An adverse event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with the treatment. A Serious Adverse Event is defined as any untoward medical occurrence that, at any dose results in death or is life-threatening or requires inpatient hospitalization
Time Frame: AEs: Day 1 to Day 11 (Part A), Day 1 to Day 24 (Part B); SAEs: Day -21 to within 30 days of discontinuation of dosing (Part A), Day -21 to within 30 days of discontinuation of dosing (Part B)
Population: All participants who had received at least one dose of BMS-986251 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 3 | 1 | 1
Participants
  % of participants that experienced SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  % of participants that died | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  % of participants with AE leading to study discon. | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Changes in Vital Signs
Description: Vital signs (Systolic and diastolic blood pressure and pulse) were recorded after the participant had been resting for at least 5 minutes in the supine position.
Time Frame: Part A: Days 1, 2, 3, 4, 5, 6, 7, 9 and 11; Part B: Days 1, 2-13, 15, 16, 18, 20, 24
Population: All participants who had received at least one dose of BMS-986251 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 3 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Changes in Electrocardiogram (ECG) Parameters
Description: The following ECG parameters were recorded: heart rate, PR-interval, QRS-duration, QT-interval, QTcinterval, (Fridericia's) and the interpretation of the ECG profile by the Investigator
Time Frame: Part A: Days 1, 2, 3,5, 7 and 11; Part B: Days 1, 2, 4, 6, 8, 10, and 12,24
Population: All participants who had received at least one dose of BMS-986251 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 3 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Changes in Clinical Laboratory Parameters
Description: Hematology: Hemoglobin, Hematocrit, Total leukocyte count, including differential Platelet count, Red blood cell count, Reticulocyte count; Chemistry:
  Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Total bilirubin, Direct bilirubin, Alkaline phosphatase, Lactate dehydrogenase , (LDH), Creatinine, Urea, Uric acid, Fasting glucose, High sensitivity C-reactive protein (hs-CRP), Total protein, Albumin Sodium, Potassium, Chloride, Calcium Inorganic phosphate, Magnesium, Creatine kinase, Creatinine clearance (CLcr)- screening only, Cholesterol Triglycerides, High-density lipoprotein (HDL), Low-density lipoprotein (LDL), Urinalysis: Protein, Glucose, Blood Leukocyte esterase, Specific gravity, pH,Microscopic examination of the sediment if blood, protein or leukocytes esterase are positive on the dipstick; Other Analyses: Urine test for alcohol, Urine test for drugs of abuse, Pregnancy test
Time Frame: Part A: Days 2, 4, 7 and 11; Part B: Days 3, 7, 10, 14, 16, 24
Population: All participants who had received at least one dose of BMS-986251 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 3 | 1 | 1
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part A: Days 1, 2, 3, 4, 5, 6, 7, 9, 11; Part B : Day 1 and 14
Population: All participants who received at least 1 dose of BMS-986251 and had any available concentration-time data. Additionally, the evaluable PK population was defined as participants who had adequate PK profiles.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 3 | 0 | 1
ng/mL |  | 74.3 (5.88) | 206 (55.8) | 659 (207) | 1131 (278) | 2147 (175) |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

6. Primary Outcome: Time of Maximum Observed Plasma Concentration (Tmax)
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part A: Days 1, 2, 3, 4, 5, 6, 7, 9, 11; Part B : Day 1 and 14
Population: as for outcome 5
Measure: Median (Full Range); unit: h
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 3 | 0 | 1
h |  | 3.50 [1.50 to 6.00] | 2.27 [1.02 to 4.02] | 1.53 [1.02 to 8.00] | 2.53 [2.02 to 4.02] | 1.05 [1.02 to 1.07] |  | NA [NA to NA] — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

7. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration [AUC(0-t)]
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part A: Days 1, 2, 3, 4, 5, 6, 7, 9, 11; Part B : Day 1 and 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 3 | 0 | 1
ng.h/mL |  | 5530 (954) | 14737 (3339) | 36318 (9554) | 71172 (13328) | 126198 (21811) |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

8. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time [AUC(0-inf)] (Part A)
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part A: Days 1, 2, 3, 4, 5, 6, 7, 9, 11
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 3
ng.h/mL |  | 6052 (1221) | 15815 (3926) | 38080 (10827) | 75335 (14726) | 130873 (24294)

9. Primary Outcome: Terminal Elimination Half-life, Calculated as 0.693/Kel [t(1/2)]
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part A: Days 1, 2, 3, 4, 5, 6, 7, 9, 11; Part B : Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 3 | 0 | 1
h |  | 70.9 (16.5) | 62.6 (15.0) | 52.2 (9.02) | 54.6 (13.6) | 48.2 (7.02) |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

10. Primary Outcome: Apparent (Oral) Clearance (CL/F) Calculated as Dose/[AUC(0-inf)] for Single Dose
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part A: Day 1, Part B: Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 3 | 0 | 1
L/h |  | 0.343 (0.076) | 0.400 (0.100) | 0.419 (0.109) | 0.411 (0.078) | 0.469 (0.083) |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

11. Primary Outcome: Apparent Volume of Distribution at Terminal Phase [V(z)/F]
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part A: Days 1, 2, 3, 4, 5, 6, 7, 9, 11; Part B : Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 3 | 0 | 1
L |  | 34.1 (6.39) | 35.3 (8.52) | 30.6 (5.54) | 32.3 (9.44) | 32.1 (3.98) |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

12. Primary Outcome: Cumulative Urinary Excretion (of the Unchanged Drug) [Ae(t)]
Description: Summary of BMS-986251 Excretion Parameters in Urine. PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part A: Days 1, 2, 3, 4, 5, 6, 7 ; Part B : Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 3 | 0 | 1
mg |  | 0 (0) | 0 (0) | 0.002 (0.002) | 0.009 (0.002) | 0.020 (0.011) |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

13. Primary Outcome: Amount Excreted Unchanged in Urine (% of Dose) [Fe(Urine)%]
Description: as for outcome 12
Time Frame: Part A: Days 1, 2, 3, 4, 5, 6, 7 ; Part B : Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of dose
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 3 | 0 | 1
Percentage of dose |  | 0 (0) | 0 (0) | 0.012 (0.011) | 0.031 (0.007) | 0.033 (0.018) |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

14. Primary Outcome: Renal Clearance [CL(R)]
Description: as for outcome 12
Time Frame: Part A: Days 1, 2, 3, 4, 5, 6, 7 ; Part B : Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 6 | 6 | 6 | 6 | 3 | 0 | 1
L/h |  | 0 (0) | 0 (0) | 0.00005 (0.00004) | 0.00016 (0.00006) | 0.00019 (0.00012) |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

15. Primary Outcome: Area Under the Concentration-time Curve Over 24 Hours (One Dosing Interval) [AUC(0-24)] (Part B)
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part B : Days 1 and Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 1
ng.h/mL |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

16. Primary Outcome: Ratio of AUC(0-24) Following Last Dose to AUC(0-24) Following First Dose [AR[AUC(0-24)]] (Part B)
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part B : Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 1
Ratio |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

17. Primary Outcome: Ratio of Cmax Following Last Dose to Cmax Following First Dose [AR(Cmax)] (Part B)
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part B : Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 1
Ratio |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

18. Primary Outcome: Pre-dose Plasma Concentration (Cpre) (Part B)
Description: PK parameters were derived from BMS-986251 concentration versus time data measured at the time points specified
Time Frame: Part B : Days 2-14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 0 | 1
ng/mL |  | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

19. Secondary Outcome: Maximum Observed Inhibition [I(Max)]
Description: Summary of IL-17 Inhibition in Whole Blood Pharmacodynamic (PD) Parameters
Time Frame: Part A: Days 1, 2, 3, 5, 7, 11 ; Part B : Day 1, 2, 16, 20, 24
Population: All participants who received at least 1 dose of BMS-986251 or placebo and had any available concentration-time data for the PD assessments. Additionally, the evaluable PD population was defined as participants who had adequate PD profiles.
Measure: Mean (Standard Deviation); unit: Percent inhibition
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 3 | 1 | 1
Percent inhibition | 27.0 (24.0) | 36.9 (9.54) | 44.2 (8.89) | 58.2 (4.18) | 72.7 (11.3) | 73.9 (10.9) | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

20. Secondary Outcome: Time of Maximum Observed Inhibition [t(Imax)]
Description: Summary of IL-17 Inhibition in Whole Blood Pharmacodynamic (PD) Parameters
Time Frame: Part A: Days 1, 2, 3, 5, 7, 11 ; Part B : Day 1, 2, 16, 20, 24
Population: as for outcome 19
Measure: Median (Full Range); unit: h
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 3 | 1 | 1
h | 2.00 [1.00 to 240.00] | 1.00 [1.00 to 24.00] | 13.00 [1.00 to 240.00] | 1.00 [1.00 to 48.00] | 1.00 [1.00 to 24.00] | 2.00 [1.00 to 4.00] | NA [NA to NA] — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality | NA [NA to NA] — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

21. Secondary Outcome: Time of Inhibition Above 50% [t(I>50%)]
Description: Summary of IL-17 Inhibition in Whole Blood Pharmacodynamic (PD) Parameters
Time Frame: Part A: Days 1, 2, 3, 5, 7, 11 ; Part B : Day 1, 2, 16, 20, 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 3 | 1 | 1
h | NA (NA) — Inhibition>50% showed an intermittent pattern (above and below 50%) over time. Due to the variation over time it was not possible to calculate a reliable [t (I>50%) | NA (NA) — Inhibition>50% showed an intermittent pattern (above and below 50%) over time. Due to the variation over time it was not possible to calculate a reliable [t (I>50%) | NA (NA) — Inhibition>50% showed an intermittent pattern (above and below 50%) over time. Due to the variation over time it was not possible to calculate a reliable [t (I>50%) | NA (NA) — Inhibition>50% showed an intermittent pattern (above and below 50%) over time. Due to the variation over time it was not possible to calculate a reliable [t (I>50%) | NA (NA) — Inhibition>50% showed an intermittent pattern (above and below 50%) over time. Due to the variation over time it was not possible to calculate a reliable [t (I>50%) | NA (NA) — Inhibition>50% showed an intermittent pattern (above and below 50%) over time. Due to the variation over time it was not possible to calculate a reliable [t (I>50%) | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

22. Secondary Outcome: Time of Inhibition Above 90% [t(I>90%)]
Description: Summary of IL-17 Inhibition in Whole Blood Pharmacodynamic (PD) Parameters
Time Frame: Part A: Days 1, 2, 3, 5, 7, 11 ; Part B : Day 1, 2, 16, 20, 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 3 | 1 | 1
h | NA (NA) — Data did not allow for these calculations | NA (NA) — Data did not allow for these calculations | NA (NA) — Data did not allow for these calculations | NA (NA) — Data did not allow for these calculations | NA (NA) — Data did not allow for these calculations | NA (NA) — Data did not allow for these calculations | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

23. Secondary Outcome: Pre-dose Inhibition [I(Pre)] (Part B)
Description: Summary of IL-17 Inhibition in Whole Blood Pharmacodynamic (PD) Parameters
Time Frame: Part B : Days 2, 4, 7, and 14
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Percent inhibition
Arm/Group | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 1 | 1
Percent inhibition | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

24. Primary Outcome: Inhibition at Time t [I(t)] (Part B)
Description: Summary of IL-17 Inhibition in Whole Blood Pharmacodynamic (PD) Parameters
Time Frame: Part B : Days 16, 20, and 24
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Percent inhibition
Arm/Group | Part B: Placebo | Part B: 3 mg QD (Once Daily)
Number analyzed (Participants) | 1 | 1
Percent inhibition | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality | NA (NA) — Due to the early termination of the study, only one subject was exposed to multiple doses of BMS-986251 in Part B.Individual data not presented to maintain confidentiality

ADVERSE EVENTS:
Time Frame: AEs: Day 1 to Day 11 (Part A), Day 1 to Day 24 (Part B); SAEs: Day -21 to within 30 days of discontinuation of dosing (Part A), Day -21 to within 30 days of discontinuation of dosing (Part B) (Approximately 9 months)
Arm/Group | Part A: Placebo | Part A: BMS-986251 2 mg | Part A: BMS-986251 6 mg | Part A: BMS-986251 15 mg | Part A: BMS-986251 30 mg | Part A : BMS-986251 60 mg | Part B: Placebo | Part B: 3 mg QD (Once Daily)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/3 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 5/9 | 4/6 | 4/6 | 5/6 | 4/6 | 3/3 | 0/1 | 0/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=9) | Part A: BMS-986251 2 mg (N=6) | Part A: BMS-986251 6 mg (N=6) | Part A: BMS-986251 15 mg (N=6) | Part A: BMS-986251 30 mg (N=6) | Part A : BMS-986251 60 mg (N=3) | Part B: Placebo (N=1) | Part B: 3 mg QD (Once Daily) (N=1)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Vessel Puncture Site Reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Catheter Site Haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter Site Related Reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Complication Associated With Device (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Medical Device Site Reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Poor Quality Sleep (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the early termination of the study, only one participant was exposed to multiple doses of BMS-986251.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03329885/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03329885/SAP_001.pdf